CLINICAL TRIAL: NCT07099729
Title: Comparison of the Dynamic Mechanical Power Formula With the Geometric Method in Volume-Controlled and Pressure-Controlled Ventilation Modes in Patients With Acute Respiratory Distress Syndrome: A Prospective Validation Study
Brief Title: Comparison of Dynamic Mechanical Power Formula With Geometric Method in Pressure- and Volume-Controlled Ventilation: A Validation Study
Status: Completed | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Furkan Tontu, Specialist Doctor, Başakşehir Çam & Sakura City Hospital
Other Study IDs: 2025-76
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS); Ventilated Patient in Intensive Care
Keywords: mechanical power; volume control ventilation; pressure control ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ARDS patients group: This group includes all patients diagnosed with Acute Respiratory Distress Syndrome (ARDS) who underwent both volume-controlled ventilation (VCV) and pressure-controlled ventilation (PCV) modes in a sequential and crossover manner.
  Interventions: Other: Volume-Controlled Ventilation (VCV) with inspiratory-to-expiratory (I:E) ratio of 1:2.; Other: Volume-Controlled Ventilation (VCV) with inspiratory-to-expiratory (I:E) ratio of 1:1.; Other: Pressure-Controlled Ventilation (PCV) with inspiratory-to-expiratory (I:E) ratio of 1:2.; Other: Pressure-Controlled Ventilation (PCV) with inspiratory-to-expiratory (I:E) ratio of 1:1.

INTERVENTIONS:
Other: Volume-Controlled Ventilation (VCV) with inspiratory-to-expiratory (I:E) ratio of 1:2. — Patients received volume-controlled ventilation (VCV) with an inspiratory-to-expiratory (I:E) ratio of 1:2. Mechanical power was calculated geometrically (MPgeo) using ventilator screenshots, and results were compared with dynamic mechanical power (MPdyn) values.
Other: Volume-Controlled Ventilation (VCV) with inspiratory-to-expiratory (I:E) ratio of 1:1. — Patients received volume-controlled ventilation (VCV) with an inspiratory-to-expiratory (I:E) ratio of 1:1. MPgeo was computed from ventilator screenshots and compared to MPdyn values to assess agreement.
Other: Pressure-Controlled Ventilation (PCV) with inspiratory-to-expiratory (I:E) ratio of 1:2. — Patients received pressure-controlled ventilation (PCV) with an I:E ratio of 1:2. Mechanical power was measured using both geometric (MPgeo) and dynamic (MPdyn) methods for validation purposes.
Other: Pressure-Controlled Ventilation (PCV) with inspiratory-to-expiratory (I:E) ratio of 1:1. — Patients received pressure-controlled ventilation (PCV) with an I:E ratio of 1:1. Geometric mechanical power calculations from ventilator screenshots were compared with MPdyn values for accuracy assessment.

SUMMARY:
This prospective observational study aims to validate the dynamic mechanical power (MPdyn) formula by comparing it with the gold-standard geometric method (MPgeo) in patients with acute respiratory distress syndrome (ARDS) who are mechanically ventilated in volume-controlled ventilation (VCV) and pressure-controlled ventilation (PCV) modes.

Mechanical power (MP) is a composite parameter that integrates multiple components of ventilator-induced lung injury (VILI) and has shown strong associations with mortality in ARDS. While several formulas exist for calculating MP in VCV and PCV modes, most require inspiratory resistance, which is not readily available at the bedside. The MPdyn formula, introduced by Asar et al., allows for bedside calculation without inspiratory resistance and has shown good agreement with established formulas such as MPrs and MPLM. However, it has never been validated against the geometric method, which calculates mechanical power based on the area of the pressure-volume (P-V) loop and is considered the most accurate standard.

In this single-center study, 37 deeply sedated ARDS patients were ventilated with a Servo-U ventilator using both VCV and PCV modes. For each mode, two different I:E ratios (1:2 and 1:1) were applied, and 12 screenshots of full P-V loops were captured per patient, totaling 444 images. Geometric MP (MPgeo) was calculated using Python-based image processing with OpenCV and NumPy libraries. Dynamic mechanical power (MPdyn) was computed using ventilator-recorded values of minute volume (MVe), work of breathing per liter (WOBv), and PEEP.

The primary outcome was the agreement between MPdyn and MPgeo values under different ventilator modes and I:E ratios. Secondary outcomes included regression correlation (R²) and Bland-Altman analysis of bias and limits of agreement. This study seeks to determine whether MPdyn is a valid and reliable surrogate for geometric mechanical power, particularly in clinical settings where bedside calculation is needed and inspiratory resistance cannot be easily measured.

DETAILED DESCRIPTION:
Mechanical power (MP) is an integrative parameter that quantifies the energy delivered to the lungs during mechanical ventilation. It accounts for multiple factors contributing to ventilator-induced lung injury (VILI), including tidal volume, airway pressures, respiratory rate, compliance, and resistance. MP has been shown to correlate strongly with morbidity and mortality in critically ill patients, particularly those with acute respiratory distress syndrome (ARDS).

Several MP calculation formulas have been proposed for volume-controlled ventilation (VCV) and pressure-controlled ventilation (PCV). While formulas such as MPrs (Gattinoni) and MPLM (Trinkle) are widely used, many of them require precise measurement of inspiratory resistance (Raw), which is often not readily accessible at the bedside-especially in PCV. To address this, a dynamic mechanical power formula (MPdyn) was developed by Asar et al., which estimates MP without the need for inspiratory resistance. MPdyn has demonstrated good agreement with MPrs in VCV and with MPLM in PCV. However, it has not been directly validated against the geometric method, which remains the gold standard for MP calculation.

The geometric method involves calculating the area enclosed by the pressure-volume (P-V) loop on the ventilator screen. This area represents the energy per breath, which can be multiplied by respiratory rate to yield MP. Modern ventilators, such as the Maquet Servo-U, provide high-resolution graphical displays that allow for precise area calculations using digital image processing.

This prospective observational study was conducted in the intensive care unit of Bakırköy Dr. Sadi Konuk Training and Research Hospital, Istanbul. A total of 37 ARDS patients who were deeply sedated and under controlled mechanical ventilation were enrolled. Each patient was ventilated in both VCV and PCV modes with two different I:E ratios (1:2 and 1:1). For each setting, three screenshots of the P-V loop were captured, resulting in 12 images per patient and 444 images in total.

Geometric mechanical power (MPgeo) was calculated using Python-based image analysis (OpenCV, NumPy, and PIL libraries). The region of interest (ROI) corresponding to the P-V loop was extracted, binarized, and segmented to compute the loop area. This pixel-based area was then scaled using the known tidal volume (TVe) and pressure (Pinsp) values to obtain mechanical energy per breath. MPgeo was calculated as:

MPgeo (J/min) = [E_breath × RR] + [PEEP × TVe × RR × 0.098]

Dynamic mechanical power (MPdyn) was calculated using the following formula:

MPdyn = MVe × [WOBv + (PEEP × 0.098)] where MVe is the expiratory minute volume (L/min), WOBv is the work of breathing per liter (J/L), and PEEP is the end-expiratory pressure (cmH₂O).

Statistical analysis included descriptive statistics, Shapiro-Wilk test for normality, univariable linear regression to assess correlation between MPdyn and MPgeo, and Bland-Altman analysis to evaluate agreement between methods. Paired measurements were analyzed both at the patient-averaged level and for all individual data points.

The primary outcome of the study was the degree of agreement between MPdyn and MPgeo under different ventilator modes (VCV, PCV) and I:E ratios (1:1, 1:2). Secondary analyses included evaluating potential biases and limits of agreement.

This study is expected to validate MPdyn as a reliable, practical alternative to geometric calculations in clinical settings, facilitating routine bedside monitoring of mechanical power without requiring complex measurements or advanced equipment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of moderate-to-severe ARDS according to the Berlin criteria
* Receiving mechanical ventilation in volume-controlled (VCV) or pressure-controlled (PCV) mode
* Stable hemodynamics during data collection
* Expected to remain under mechanical ventilation for at least 48 hours
* Written informed consent from legal representative

Exclusion Criteria:

* Presence of chest tube or pneumothorax
* Known neuromuscular disease affecting respiratory function
* Pregnancy
* Patients with do-not-resuscitate (DNR) or limitation-of-therapy orders
* Incomplete ventilator data or poor-quality screenshots

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult ICU patients diagnosed with ARDS and receiving mechanical ventilation (VCV or PCV mode) at a tertiary care hospital. Data will be collected between 24 and 48 hours after ICU admission.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Agreement Between Dynamic Mechanical Power (MPdyn) and Geometric Mechanical Power (MPgeo) Across Ventilation Modes and I:E Ratios | Between 24 and 48 hours after ICU admission
  To assess the agreement between MPdyn (calculated using the dynamic mechanical power formula) and MPgeo (calculated from ventilator screenshots) in patients with ARDS under four different ventilation settings:
  VCV with I:E 1:2 VCV with I:E 1:1 PCV with I:E 1:2 PCV with I:E 1:1 Agreement will be quantified using Bland-Altman analysis and correlation coefficients.

CONTACTS AND LOCATIONS:
Locations (1):
- Bakirkoy Sadi Konuk Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared due to institutional restrictions and ethical considerations concerning patient confidentiality.

REFERENCES:
- [Background] Marini JJ, Rodriguez RM, Lamb V. Bedside estimation of the inspiratory work of breathing during mechanical ventilation. Chest. 1986 Jan;89(1):56-63. doi: 10.1378/chest.89.1.56. PMID 3940790
- [Background] Cabello B, Mancebo J. Work of breathing. Intensive Care Med. 2006 Sep;32(9):1311-4. doi: 10.1007/s00134-006-0278-3. Epub 2006 Jul 13. No abstract available. PMID 16838150
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] Acicbe O, Ozgur CY, Rahimi P, Canan E, Asar S, Cukurova Z. The effect of inspiratory rise time on mechanical power calculations in pressure control ventilation: dynamic approach. Intensive Care Med Exp. 2023 Dec 20;11(1):98. doi: 10.1186/s40635-023-00584-6. PMID 38117345
- [Background] Iotti GA, Braschi A, Brunner JX, Smits T, Olivei M, Palo A, Veronesi R. Respiratory mechanics by least squares fitting in mechanically ventilated patients: applications during paralysis and during pressure support ventilation. Intensive Care Med. 1995 May;21(5):406-13. doi: 10.1007/BF01707409. PMID 7665750
- [Background] Asar S, Acicbe O, Sabaz MS, Kucur Tulubas E, Hergunsel GO, Cukurova Z, Canan E, Cakar N. Simplified calculation of mechanical power for pressure controlled ventilation in Covid-19 ARDS patients. Minerva Anestesiol. 2022 Jan-Feb;88(1-2):42-50. doi: 10.23736/S0375-9393.21.15741-4. PMID 35224956
- [Background] van der Meijden S, Molenaar M, Somhorst P, Schoe A. Calculating mechanical power for pressure-controlled ventilation. Intensive Care Med. 2019 Oct;45(10):1495-1497. doi: 10.1007/s00134-019-05698-8. Epub 2019 Jul 29. No abstract available. PMID 31359082
- [Background] Becher T, van der Staay M, Schadler D, Frerichs I, Weiler N. Calculation of mechanical power for pressure-controlled ventilation. Intensive Care Med. 2019 Sep;45(9):1321-1323. doi: 10.1007/s00134-019-05636-8. Epub 2019 May 17. No abstract available. PMID 31101961
- [Background] Chi Y, He H, Long Y. A simple method of mechanical power calculation: using mean airway pressure to replace plateau pressure. J Clin Monit Comput. 2021 Oct;35(5):1139-1147. doi: 10.1007/s10877-020-00575-y. Epub 2020 Aug 11. PMID 32780353
- [Background] Giosa L, Busana M, Pasticci I, Bonifazi M, Macri MM, Romitti F, Vassalli F, Chiumello D, Quintel M, Marini JJ, Gattinoni L. Mechanical power at a glance: a simple surrogate for volume-controlled ventilation. Intensive Care Med Exp. 2019 Nov 27;7(1):61. doi: 10.1186/s40635-019-0276-8. PMID 31773328
- [Background] Asar S, Acicbe O, Cukurova Z, Hergunsel GO, Canan E, Cakar N. Bedside dynamic calculation of mechanical power: A validation study. J Crit Care. 2020 Apr;56:167-170. doi: 10.1016/j.jcrc.2019.12.027. Epub 2020 Jan 2. PMID 31931417
- [Background] Serpa Neto A, Deliberato RO, Johnson AEW, Bos LD, Amorim P, Pereira SM, Cazati DC, Cordioli RL, Correa TD, Pollard TJ, Schettino GPP, Timenetsky KT, Celi LA, Pelosi P, Gama de Abreu M, Schultz MJ; PROVE Network Investigators. Mechanical power of ventilation is associated with mortality in critically ill patients: an analysis of patients in two observational cohorts. Intensive Care Med. 2018 Nov;44(11):1914-1922. doi: 10.1007/s00134-018-5375-6. Epub 2018 Oct 5. PMID 30291378
- [Background] Gattinoni L, Tonetti T, Cressoni M, Cadringher P, Herrmann P, Moerer O, Protti A, Gotti M, Chiurazzi C, Carlesso E, Chiumello D, Quintel M. Ventilator-related causes of lung injury: the mechanical power. Intensive Care Med. 2016 Oct;42(10):1567-1575. doi: 10.1007/s00134-016-4505-2. Epub 2016 Sep 12. PMID 27620287
- [Background] Trinkle CA, Broaddus RN, Sturgill JL, Waters CM, Morris PE. Simple, accurate calculation of mechanical power in pressure controlled ventilation (PCV). Intensive Care Med Exp. 2022 May 30;10(1):22. doi: 10.1186/s40635-022-00448-5. PMID 35644896